CLINICAL TRIAL: NCT02537925
Title: The Effect of Celecoxib on Concurrent Chemoradiation With Weekly Nedaplatin in Nasopharyngeal Carcinoma
Brief Title: The Effect of COX-2 Inhibitor on Radiosensitivity in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changjie Huang (Other)
Responsible Party: Sponsor-Investigator, Changjie Huang, head of the medical department, Nanning Second People's Hospital
Organization: Nanning Second People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NaningSPH_2014
Record Dates: First submitted 2015-05-17; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: COX-2 inhibitors; radiosensitivity; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Celecoxib; Cyclooxygenase 2 Inhibitors; nedaplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- concurrent_radiochemotherapy (Active Comparator): Concurrent radiotherapy with Nedaplatin 40mg/m2/week through intravenous infusion.
  Interventions: Drug: Nedaplatin; Radiation: Concurrent Radiotherapy
- celecoxib_radiochemotherapy (Experimental): Celecoxib 200mg bid po; Concurrent radiotherapy with Nedaplatin 40mg/m2/week through intravenous infusion.
  Interventions: Drug: Celecoxib; Drug: Nedaplatin; Radiation: Concurrent Radiotherapy

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 200mg bid po, to the end of concurrent radiotherapy
  Other Names: COX-2 inhibitor
  Arms: celecoxib_radiochemotherapy
Drug: Nedaplatin — 40 mg/m2, IV (in the vein) on day 1 of each 7 day cycle. Number of Cycles: to the end of concurrent radiotherapy
Radiation: Concurrent Radiotherapy — The standard radiotherapy schedules were available as conventional radiotherapy and Intensity Modulated Radiotherapy (IMRT). The cumulative radiation dose was 68~74 Gy for primary tumor (2.0~2.3 Gy/f/day, 5 day/ week, /6~7 weeks), and 50~54 Gy for lymphatic positive area (1.8 ~ 2 Gy/f/day, 5 day/week, /5.0~5.5 weeks).
  Other Names: standard radiotherapy schedule

SUMMARY:
The purpose of this study is to determine whether celecoxib is effective in the treatment of nasopharyngeal carcinoma by concurrent chemoradiation with weekly nedaplatin.

DETAILED DESCRIPTION:
1. Study Patients:

   Patients are all recruited from the Third Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China. All the patients provide written informed consent before enrollment. All eligible patients received a pretreatment evaluation including complete history and physical examination, endoscopic biopsy, routine laboratory tests for hematologic, renal and hepatic function as well as a dental and nutritional evaluation prior to treatment. Radiological investigations consisted of computed tomography (CT) scan or magnetic MRI of the nasopharynx, chest radiography, ultrasound of the upper abdomen and bone scintigraphy. Pathologic confirmation of nasopharyngeal cancer (NPC) was performed and re-classified according to the world health organization (WHO) subtypes.
2. Study design:

   A total of 120 NPC patients are randomly and equally divided into two groups: Nedaplatin alone concurrent radiotherapy, Celecoxib plus nedaplatin concurrent radiotherapy. The tumor response will be evaluated by magnetic resonance imaging (MRI) after 4 weeks. The tumor responses including Complete Response (CR), Partial Response (PR) , Stable Disease (SD) and Progressive Disease (PD) is defined according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0. The show term or long term toxicity will be evaluated according to the National Cancer Institute Common Toxicity Criteria (NCICTC), version 3.0. All the NPC patients are requested to be followed up with an expected average of every 3 months after the therapy.The other clinical outcomes including the first evidence of cancer progression or death from any cause, the occurrence of distant metastasis, and the relapse of a local or nodal tumor will be evaluated as well. The follow-up will be up to 2018.
3. Statistical Analysis:

Statistical Package for the Social Sciences (SPSS 13.0) is used to analyze the effect of celecoxib on the nedaplatin concurrent radiotherapy. Cox's regression model and Kaplan-Meier method is used to conduct survival analysis. Clinical outcomes including the tumor responses, 1-year/3-year/5-year overall survival (OS), progression free survival (PFS), distant metastasis failure-free survival (DMFS) and locoregional failure-free survival (LFFS) will be analyzed. The multivariate Cox's regression model is used to adjust the confounders, including age and body mass index. P value less than 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Patients with NPC newly diagnosed by histopathology, and without radiotherapy or chemotherapy before the clinical trial
* Patients with measurable lesions by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* With the Eastern Cooperative Oncology Group Performance Status (ECOG PS) as 0-1 score
* Serum hemoglobin ≥10gm/dL, platelet ≥100000/μL, neutrophil granulocyte absolute counting is 1500/μL
* Serum creatinine ≤1.25 times of upper normal limit (UNL), creatinine clearance rate ≥ 60 ml/min
* Serum bilirubin ≤ 1.5times of UNL, serum aspartate aminotransferase (AST) or glutamic-oxaloacetic transaminase(GOT)≤ 2.5 times of UNL, serum alanine aminotransferase (ALT) or glutamic-pyruvic transaminase (GPT) ≤ 2.5 times of UNL, alkaline phosphatase≤5 times of UNL
* The estimate overall survival (OS)> 6 months
* With formal informed consent forms signed.

Exclusion criteria:

* With symptomatic brain/bone metastases,
* With cognitive impairment or other malignancies
* With any contraindications for radiotherapy and chemotherapy (such as active phase of infection, myocardial infarction within 6 months, symptomatic heart disease, including unstable angina pectoris, congestive heart failure or uncontrolled arrhythmias, in current immunosuppressive therapy)
* Current pregnancy, lactating women or women with fertility but don't take contraceptive measures yet
* With severe bone marrow dysfunction
* With bleeding tendency
* With abuse of drugs or alcohol addicts
* Who may have III-IV type of allergic reactions to any treatment in this study
* With termination of trial because of intolerable toxicity, other study drugs using during the clinical study, or unwilling to continue the treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with different tumor response and short term toxicity will be recorded | Patients are asked to be followed within an expected average of 4 weeks after therapy
  The tumor responses including Complete Response (CR), Partial Response (PR) , Stable Disease (SD) and Progressive Disease (PD) were evaluated by MRI, according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0; Short term toxicity was evaluated according to the National Cancer Institute Common Toxicity Criteria (NCICTC), version 3.0.

SECONDARY OUTCOMES:
The date when each patient is dead will be recorded. | Patients will be asked to be followed in an expected average of every 3 months after therapy. From date of treatment initiation until the date of first documented death from any cause, assessed up to 36 months.
  Overall survival (OS) is defined as the time between treatment initiation and the patient death.
The date when each patient shows the first evidence of cancer progression or death from any cause will be recorded. | Patients will be asked to be followed in an expected average of every 3 months after therapy. From date of treatment initiation until the date of first documented progression or date of death from any cause, whichever comes first, up to 36 months
  Progression free survival (PFS) is defined as the time between treatment initiation and the first evidence of cancer progression or death from any cause.
The date when each patient presents the occurrence of distant metastasis will be recorded. | Patients will be asked to be followed in an expected average of every 3 months after therapy. From date of treatment initiation until the date of first documented occurrence of distant metastasis, assessed up to 36 months
  Distant metastasis failure-free survival (DMFS) is defined as the time between treatment initiation and the occurrence of distant metastasis.
The date when each patient presents the relapse of a local or nodal tumor will be recorded. | Patients will be asked to be followed in an expected average of every 3 months after therapy. From date of treatment initiation until the date of first documented relapse of a local or nodal tumor, whichever came first, assessed up to 36 months.
  Locoregional failure-free survival (LFFS) is defined as the time between treatment initiation and the relapse of a local or nodal tumor.
Long term toxicity will be recorded as the Number of Participants with Treatment-Related Adverse Events | Patients will be asked to be followed in an expected average of every 3 months after therapy. From date of treatment initiation until the documented date of the Treatment-Related Adverse Events, whichever comes first, assessed up to 36 months.
  The Treatment-Related Adverse Events are assessed by the National Cancer Institute Common Toxicity Criteria (NCICTC), version 3.0.
Age will be recorded when the therapy starts | Patients are asked to provide the birthday before the start of therapy
  Age is defined as the time between the birthday and treatment initiation.
Height in meters and weight in kilograms will be recorded when therapy starts | Patients are asked to be measured the height and weight before the start of therapy
  High and weight are measured in standing posture without shoes by trained nurses. Body mass index is calculated form weight in kilograms divided by height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: Changjie Huang, Principal Investigator — The third Affiliated Hospital of Guangxi Medical University
Locations (1):
- The third Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Background] Soo RA, Wu J, Aggarwal A, Tao Q, Hsieh W, Putti T, Tan KB, Low JS, Lai YF, Mow B, Hsu S, Loh KS, Tan L, Tan P, Goh BC. Celecoxib reduces microvessel density in patients treated with nasopharyngeal carcinoma and induces changes in gene expression. Ann Oncol. 2006 Nov;17(11):1625-30. doi: 10.1093/annonc/mdl283. Epub 2006 Sep 28. PMID 17008411
- [Background] Mohammadianpanah M, Razmjou-Ghalaei S, Shafizad A, Ashouri-Taziani Y, Khademi B, Ahmadloo N, Ansari M, Omidvari S, Mosalaei A, Mosleh-Shirazi MA. Efficacy and safety of concurrent chemoradiation with weekly cisplatin +/- low-dose celecoxib in locally advanced undifferentiated nasopharyngeal carcinoma: a phase II-III clinical trial. J Cancer Res Ther. 2011 Oct-Dec;7(4):442-7. doi: 10.4103/0973-1482.92013. PMID 22269407